CLINICAL TRIAL: NCT00608582
Title: Transcranial Magnetic Stimulation to Improve Speech
Brief Title: Transcranial Magnetic Stimulation to Improve Speech in Aphasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Harvard Medical School (HMS and HSDM) (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Margaret Naeser, Research Professor of Neurology, Boston University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NIH-DC05672; R01DC005672 (NIH); Boston Medical Ctr IRB-H22484 (Other: Boston University School of Medicine); VA Boston Healthcare IRB-1145 (Other: VA Boston Healthcare System)
Record Dates: First submitted 2008-01-24; First posted 2008-02-06 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Aphasia; Cerebrovascular Stroke
Keywords: Transcranial Magnetic Stimulation, Repetitive; TMS; Treat Naming; Aphasia; Chronic Stroke; Randomized, Controlled Trial
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real rTMS (Experimental): These patients receive a series of 10 Real Transcranial Magnetic Stimulation, Repetitive (rTMS), treatments, only. There is pre-testing, and post-testing at 2 months after the last Real rTMS treatment.
  Interventions: Device: Transcranial Magnetic Stimulation, Repetitive
- Sham rTMS (Sham Comparator): Patients receive a series of 10 Sham Transcranial Magnetic Stimulation, Repetitive (rTMS) treatments, followed by a series of 10 Real rTMS treatments. Sham rTMS treatments are identical to the Real rTMS treatments, however, no magnetic pulse is released. There is pre-testing, and post-testing at 2 months after the last Sham rTMS treatment.
  Interventions: Device: Transcranial Magnetic Stimulation, Repetitive

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation, Repetitive — 10 rTMS treatments (90% of motor threshold, 20 minutes, at 1 Hz) to specific right hemisphere area of brain cortex; 5 days per week for 2 weeks at the Berenson-Allen Center for Noninvasive Brain Stimulation, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, MA; or at the Neurology Department, Hospital of the University of Pennsylvania, Philadelphia, PA.

SUMMARY:
The purpose of this study is to examine whether repetitive transcranial magnetic stimulation (rTMS) can be used to improve speech in chronic stroke patients with aphasia. Aphasia patients can have problems with speech production. The rTMS procedure allows painless, noninvasive stimulation of human cortex from outside the head.

Chronic aphasia patients have been observed in our functional magnetic resonance brain imaging studies to have excess brain activation in brain areas possibly related to language on the right side of the brain (opposite side to where the stroke took place). It is expected that suppression of activity in the directly targeted brain region will have an overall modulating effect on the neural network for naming (and propositional speech) and will result in behavioral improvement.

DETAILED DESCRIPTION:
OBJECTIVE: The purpose of this research is to investigate whether repetitive transcranial magnetic stimulation (rTMS) can improve speech in chronic stroke patients with aphasia. TMS allows painless, noninvasive stimulation of brain cortex (1 cm x 1 cm). Slow (1 Hz) rTMS appears to decrease excitability in the targeted cortical region of interest (ROI) leading to measurable behavioral effects. Chronic aphasia patients have been observed in our fMRI work (and others) to have increased activation in right (R) Broca's and other R language homologues during language tasks. It is hypothesized that suppression of activity in a directly targeted right hemisphere (RH) ROI will have an overall modulating effect on functionally connected elements of the distributed neural network for naming (and propositional speech), and will result in behavioral improvement.

RESEARCH PLAN AND METHODS:

Nonfluent aphasia patients (>6 Mo. poststroke) will be studied. The rTMS treatments in Boston take place at the Berenson-Allen Center for Noninvasive Brain Stimulation, Beth Israel Deaconess Medical Center, Harvard Medical School under the supervision of Alvaro Pascual-Leone, M.D., Ph.D. and additional patients will be studied at the Hospital of the University of Pennsylvania, H. Branch Coslett, M.D., who is a P.I. on that subcontract. This is a blinded, randomized, sham-control, incomplete crossover design. Naming and language tests are obtained pre- and post- rTMS.

Treatment Design: Multiple Baseline Language Evaluations (x3) are performed at Entry (Boston Naming Test, BNT; and Boston Diagnostic Aphasia Exam, BDAE). Primary Outcome Measures are BNT; and Number of Words per Longest Phrase Length (cookie theft picture description) from the BDAE. Patients are randomly assigned to receive a series of either Sham rTMS followed by a series of Real rTMS; OR they receive only the series of Real rTMS. The Sham series is identical to the Real, however, no magnetic pulse is emitted from the coil, although the patient hears the same clicking sound emitted from the coil. Due to space limitation here, only the Real rTMS treatment schedule is described.

There are two rTMS Phases: During Phase 1, the single, best RH cortical ROI to suppress with rTMS to improve picture naming, is determined for each patient. Real rTMS (1 Hz, 90% motor threshold) is applied for 10 minutes, in separate rTMS sessions, to each of 4 different RH cortical ROIs (R ant. BA 45; R post. BA 45; R BA 44 and R M1, mouth). Snodgrass & Vanderwart (S&V, 1980) Picture Naming is tested immediately before and after each ROI has been suppressed with rTMS. The single RH ROI which is associated with at least a 2 SD improvement (above S&V Naming, tested 3x at Baseline), immediately following 10 minutes of rTMS to suppress that cortical area, is considered to be the Best Response ROI for that patient. During Phase 2, the Best Response ROI from Phase 1 is suppressed for 20 minutes, 5 days per week, 2 weeks. All patients receive follow-up BNT and BDAE testing at 2 months following the 10th Real (or Sham) rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Right Handed
* Single, Left Hemisphere Cerebrovascular Stroke
* Must be at least 6 months poststroke onset
* Native Speaker of English
* Clinical Diagnosis of Aphasia

Exclusion Criteria:

* Intracranial metallic body from prior neurosurgical procedure
* Implanted metallic devices: pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit or ventriculoperitoneal shunt
* Past history of seizure within 1 year
* Pregnancy
* History of substance abuse within last 6 months

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2002-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Naeser, Ph.D., Study Chair — Department of Neurology, Boston University School of Medicine, Boston, MA; H B Coslett, M.D., Principal Investigator — Department of Neurology, Hospital of the University of Pennsylvania, Philadelphia, PA; Alvaro Pascual-Leone, M.D., Ph.D., Principal Investigator — Berenson-Allen Center for Noninvasive Brain Stimulation, Department of Neurology, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, MA
Locations (3):
- United States (3):
  - VA Boston Healthcare System, Jamaica Plain Campus, Boston University Aphasia Research Center (12-A), 150 So. Huntington Ave., Boston, Massachusetts
  - Berenson-Allen Center for Noninvasive Brain Stimulation, 330 Brookline Ave, Kirstein Bldg., Dept. of Neurology, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts
  - Department of Neurology, Hospital of the University of Pennsylvania, 3 W. Gates Bldg., Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin PI, Naeser MA, Ho M, Treglia E, Kaplan E, Baker EH, Pascual-Leone A. Research with transcranial magnetic stimulation in the treatment of aphasia. Curr Neurol Neurosci Rep. 2009 Nov;9(6):451-8. doi: 10.1007/s11910-009-0067-9. PMID 19818232
- [Background] Naeser MA, Martin PI, Treglia E, Ho M, Kaplan E, Bashir S, Hamilton R, Coslett HB, Pascual-Leone A. Research with rTMS in the treatment of aphasia. Restor Neurol Neurosci. 2010;28(4):511-29. doi: 10.3233/RNN-2010-0559. PMID 20714075
- [Background] Hamilton RH, Chrysikou EG, Coslett B. Mechanisms of aphasia recovery after stroke and the role of noninvasive brain stimulation. Brain Lang. 2011 Jul;118(1-2):40-50. doi: 10.1016/j.bandl.2011.02.005. Epub 2011 Apr 2. PMID 21459427
- [Background] Chrysikou EG, Hamilton RH. Noninvasive brain stimulation in the treatment of aphasia: exploring interhemispheric relationships and their implications for neurorehabilitation. Restor Neurol Neurosci. 2011;29(6):375-94. doi: 10.3233/RNN-2011-0610. PMID 22124035
- [Background] Naeser MA, Martin PI, Ho M, Treglia E, Kaplan E, Bashir S, Pascual-Leone A. Transcranial magnetic stimulation and aphasia rehabilitation. Arch Phys Med Rehabil. 2012 Jan;93(1 Suppl):S26-34. doi: 10.1016/j.apmr.2011.04.026. PMID 22202188
- [Background] Torres J, Drebing D, Hamilton R. TMS and tDCS in post-stroke aphasia: Integrating novel treatment approaches with mechanisms of plasticity. Restor Neurol Neurosci. 2013;31(4):501-15. doi: 10.3233/RNN-130314. PMID 23719561
- [Background] Garcia G, Norise C, Faseyitan O, Naeser MA, Hamilton RH. Utilizing repetitive transcranial magnetic stimulation to improve language function in stroke patients with chronic non-fluent aphasia. J Vis Exp. 2013 Jul 2;(77):e50228. doi: 10.3791/50228. PMID 23852365
- [Background] Naeser MA, Martin PI, Ho M, Treglia E, Kaplan E, Baker EH, and Pascual-Leone A. Transcranial Magnetic Stimulation and Aphasia Research. Book Chapter, Advances in the Neural Substrates of Language: Toward a Synthesis of Basic Science and Clinical Research. Vol 2: Language Processing in the Brain: Special Populations. Miriam Faust (Ed.), Malden, MA: Wiley-Blackwell, 2012.
- [Result] Martin PI, Naeser MA, Theoret H, Tormos JM, Nicholas M, Kurland J, Fregni F, Seekins H, Doron K, Pascual-Leone A. Transcranial magnetic stimulation as a complementary treatment for aphasia. Semin Speech Lang. 2004 May;25(2):181-91. doi: 10.1055/s-2004-825654. PMID 15118944
- [Result] Naeser MA, Martin PI, Nicholas M, Baker EH, Seekins H, Kobayashi M, Theoret H, Fregni F, Maria-Tormos J, Kurland J, Doron KW, Pascual-Leone A. Improved picture naming in chronic aphasia after TMS to part of right Broca's area: an open-protocol study. Brain Lang. 2005 Apr;93(1):95-105. doi: 10.1016/j.bandl.2004.08.004. PMID 15766771
- [Result] Naeser MA, Martin PI, Nicholas M, Baker EH, Seekins H, Helm-Estabrooks N, Cayer-Meade C, Kobayashi M, Theoret H, Fregni F, Tormos JM, Kurland J, Doron KW, Pascual-Leone A. Improved naming after TMS treatments in a chronic, global aphasia patient--case report. Neurocase. 2005 Jun;11(3):182-93. doi: 10.1080/13554790590944663. PMID 16006338
- [Result] Martin PI, Naeser MA, Ho M, Doron KW, Kurland J, Kaplan J, Wang Y, Nicholas M, Baker EH, Alonso M, Fregni F, Pascual-Leone A. Overt naming fMRI pre- and post-TMS: Two nonfluent aphasia patients, with and without improved naming post-TMS. Brain Lang. 2009 Oct;111(1):20-35. doi: 10.1016/j.bandl.2009.07.007. Epub 2009 Aug 19. PMID 19695692
- [Result] Naeser MA, Martin PI, Lundgren K, Klein R, Kaplan J, Treglia E, Ho M, Nicholas M, Alonso M, Pascual-Leone A. Improved language in a chronic nonfluent aphasia patient after treatment with CPAP and TMS. Cogn Behav Neurol. 2010 Mar;23(1):29-38. doi: 10.1097/WNN.0b013e3181bf2d20. PMID 20299861
- [Result] Hamilton RH, Sanders L, Benson J, Faseyitan O, Norise C, Naeser M, Martin P, Coslett HB. Stimulating conversation: enhancement of elicited propositional speech in a patient with chronic non-fluent aphasia following transcranial magnetic stimulation. Brain Lang. 2010 Apr;113(1):45-50. doi: 10.1016/j.bandl.2010.01.001. Epub 2010 Feb 16. PMID 20159655
- [Result] Naeser MA, Martin PI, Theoret H, Kobayashi M, Fregni F, Nicholas M, Tormos JM, Steven MS, Baker EH, Pascual-Leone A. TMS suppression of right pars triangularis, but not pars opercularis, improves naming in aphasia. Brain Lang. 2011 Dec;119(3):206-13. doi: 10.1016/j.bandl.2011.07.005. Epub 2011 Aug 23. PMID 21864891
- [Result] Turkeltaub PE, Coslett HB, Thomas AL, Faseyitan O, Benson J, Norise C, Hamilton RH. The right hemisphere is not unitary in its role in aphasia recovery. Cortex. 2012 Oct;48(9):1179-86. doi: 10.1016/j.cortex.2011.06.010. Epub 2011 Jun 30. PMID 21794852
- [Result] Medina J, Norise C, Faseyitan O, Coslett HB, Turkeltaub PE, Hamilton RH. Finding the Right Words: Transcranial Magnetic Stimulation Improves Discourse Productivity in Non-fluent Aphasia After Stroke. Aphasiology. 2012 Sep 1;26(9):1153-1168. doi: 10.1080/02687038.2012.710316. Epub 2012 Aug 29. PMID 23280015
- [Derived] Harvey DY, Podell J, Turkeltaub PE, Faseyitan O, Coslett HB, Hamilton RH. Functional Reorganization of Right Prefrontal Cortex Underlies Sustained Naming Improvements in Chronic Aphasia via Repetitive Transcranial Magnetic Stimulation. Cogn Behav Neurol. 2017 Dec;30(4):133-144. doi: 10.1097/WNN.0000000000000141. PMID 29256908
- See also: Aphasia Research Lab of Margaret A. Naeser, Ph.D., VA Boston Healthcare System and Dept. of Neurology, Boston University School of Medicine, Boston, MA — http://www.bu.edu/naeser/aphasia
- See also: Berenson-Allen Center for Noninvasive Brain Stimulation, Beth Israel Deaconess Medical Center, Dept. of Neurology, Harvard Medical School, Boston, MA — http://tmslab.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2002-March 2013. Recruited in hospital setting and outreach with affiliated and local clinics VA Boston Healthcare System, Boston, MA; Hospital of the University of Pennsylvania, Philadelphia, PA
Pre-assignment Details: Assessed for eligibility by telephone screen, or in-office visit. Assessment included review of medical history. Total Excluded (n = 38) Not meeting inclusion criteria (n = 31) Declined to participate (n = 2) Other reasons (n = 5)
Groups:
- Real rTMS: These patients receive a series of 10 Real rTMS treatments, only. There is pre-testing, and post-testing at 2 months after the last Real rTMS treatment.
  Transcranial Magnetic Stimulation, Repetitive: 10 rTMS treatments (90% of motor threshold, 20 minutes, at 1 Hz) to specific right hemisphere area of brain cortex; 5 days per week for 2 weeks at the Berenson-Allen Center for Noninvasive Brain Stimulation, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, MA; or at the Neurology Department, Hospital of the University of Pennsylvania, Philadelphia, PA.
- Sham rTMS: These patients receive a series of 10 Sham rTMS treatments, which are identical to the Real rTMS treatments. However, no magnetic pulse is emitted from the coil.
  There is pre-testing, and post-testing at 2 months after the last Sham rTMS treatment.
  The patients then receive a series of 10 Real rTMS treatments.
  Transcranial Magnetic Stimulation, Repetitive: 10 rTMS treatments (90% of motor threshold, 20 minutes, at 1 Hz) to specific right hemisphere area of brain cortex; 5 days per week for 2 weeks at the Berenson-Allen Center for Noninvasive Brain Stimulation, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, MA; or at the Neurology Department, Hospital of the University of Pennsylvania, Philadelphia, PA.
Period: Overall Study
Arm/Group | Real rTMS | Sham rTMS
Started | 14 | 11
Completed | 10 | 7
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — No Best Response in Phase 1 located | 1 | 1
Not completed — Illicit Drug Use | 1 | 0
Not completed — Early stage Design Change | 0 | 3

BASELINE CHARACTERISTICS:
Population: Number of participants randomized to each treatment arm
Groups:
- Sham rTMS: These patients receive a series of 10 Sham rTMS treatments, which are identical to the Real rTMS treatments. However, no magnetic pulse is emitted from the coil.
  The patients then receive a series of 10 Real rTMS treatments. There is pre-testing, and post-testing at 2 months after the last Real rTMS treatment.
  Transcranial Magnetic Stimulation, Repetitive: 10 rTMS treatments (90% of motor threshold, 20 minutes, at 1 Hz) to specific right hemisphere area of brain cortex; 5 days per week for 2 weeks at the Berenson-Allen Center for Noninvasive Brain Stimulation, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, MA; or at the Neurology Department, Hospital of the University of Pennsylvania, Philadelphia, PA.
- Total: Total of all reporting groups
Arm/Group | Real rTMS | Sham rTMS | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (7.6) | 60.8 (11) | 59.28 (9.1)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 10 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 11 | 25
Months Poststroke Onset [Mean (Standard Deviation); unit: months] — Number of months at entry after stroke
  months | 66 (40) | 51 (37) | 59 (39)

OUTCOME MEASURES:

1. Primary Outcome: Picture Naming
Description: Pictures named correctly on Boston Naming Test (BNT), First 20 Pictures
Time Frame: Baseline and 2 months after the last rTMS treatment session
Population: Chronic Stroke Patients with Aphasia who receive either a Real rTMS series or a Sham rTMS series
Measure: Mean (Standard Deviation); unit: number of pictures
Groups:
- Real rTMS: These patients receive a series of 10 Real Transcranial Magnetic Stimulation, Repetitive (rTMS) , treatments, only. There is pre-testing and post-testing at 2 months after the last Real rTMS treatment.
  Transcranial Magnetic Stimulation, Repetitive: 10 rTMS treatments (90% of motor threshold, 20 minutes, at 1 Hz) to specific right hemisphere area of brain cortex; 5 days per week for 2 weeks at the Berenson-Allen Center for Noninvasive Brain Stimulation, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, MA; or at the Neurology Department, Hospital of the University of Pennsylvania, Philadelphia, PA.
- Sham rTMS: Patients receive a series of 10 Sham Transcranial Magnetic Stimulation, Repetitive (rTMS) treatments, followed by a series of 10 Real rTMS treatments. Sham rTMS are identical to the Real rTMS treatments only no magnetic pulse is released. There is pre-testing, and post-testing at 2 months after the last Real rTMS treatment.
Arm/Group | Real rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 7
number of pictures
  Baseline | 10.3 (6.11) | 12.57 (5.88)
  2 Mo. Post rTMS | 12.1 (5.55) | 11.14 (3.24)
Statistical Analysis 1: Comparison: Real rTMS vs Sham rTMS; A repeated measures ANOVA is performed with a significance level of p<0.05 (two-sided). Factors: Time (Baseline vs. 2 Mo. Post rTMS treatment) and Group (Real vs. Sham); Test type: Superiority or Other; p < 0.028, ANOVA — p<0.05 considered significant; Post-hoc paired t-tests were performed
Statistical Analysis 2: Comparison: Real rTMS; Paired, t-tests were performed if the ANOVA yields a significant interaction (p<0.05, two-sided) for Baseline vs. 2 months after last rTMS treatment; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — p<.05 considered significant; Pairwise comparisons not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Sham rTMS; Paired, t-tests were performed if the ANOVA yields a significant interaction (p<0.05, two-sided) for Baseline vs. 2 Mo. after last Sham rTMS treatment; Test type: Superiority or Other; p < 0.237, t-test, 2 sided — p<0.05 considered significant. Pairwise comparisons were not corrected for multiple comparisons

2. Primary Outcome: Phrase Length
Description: Longest Number of Words per Phrase Length, for elicited propositional speech for BDAE Cookie Theft Picture Description
Time Frame: Baseline and 2 months after the last rTMS treatment session
Population: Chronic Stroke Patients with Aphasia who received either Real rTMS or Sham rTMS
Measure: Mean (Standard Deviation); unit: number of words per phrase length
Arm/Group | Real rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 7
number of words per phrase length
  Baseline | 5.2 (3.05) | 5.285 (3.35)
  2 Mo. Post rTMS | 5.7 (3.02) | 5.0 (3.0)
Statistical Analysis 1: Comparison: Real rTMS vs Sham rTMS; A repeated measures ANOVA is performed with a significance level of p<0.05 (two-sided). Factors: Time (Baseline vs. 2 months after last rTMS treatment) and Group (Real vs. Sham); Test type: Superiority or Other; p = 0.414, ANOVA — p<0.05 considered significant
Statistical Analysis 2: Comparison: Real rTMS vs Sham rTMS; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.822, ANOVA — p<0.05 considered significant
Statistical Analysis 3: Comparison: Real rTMS vs Sham rTMS; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.835, ANOVA — p<0.05 considered significant

ADVERSE EVENTS:
Time Frame: Through entire study period for each participant, up to 1 year
Groups:
- Real rTMS: These patients receive a series of 10 Real Transcranial Magnetic Stimulation, Repetitive (rTMS) , treatments, only. There is pre-testing, and post-testing at 2 months after the last Real rTMS treatment.
  Transcranial Magnetic Stimulation, Repetitive: 10 rTMS treatments (90% of motor threshold, 20 minutes, at 1 Hz) to specific right hemisphere area of brain cortex; 5 days per week for 2 weeks at the Berenson-Allen Center for Noninvasive Brain Stimulation, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, MA; or at the Neurology Department, Hospital of the University of Pennsylvania, Philadelphia, PA.
- Sham rTMS: Patients receive a series of 10 Sham Transcranial Magnetic Stimulation, Repetitive (rTMS) treatments, followed by a series of 10 Real rTMS treatments. There is pre-testing, and post-testing at 2 months after the last Sham rTMS treatment. Sham rTMS are identical to the Real rTMS treatments only no magnetic pulse is released. There is pre-testing, and post-testing at 2 months after the last Real rTMS treatment.
Arm/Group | Real rTMS | Sham rTMS
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No